CLINICAL TRIAL: NCT05151029
Title: The Role of Real Time Elastography in the Evaluation of Major Salivary Gland Lesions
Brief Title: Elastography in the Evaluation of Major Salivary Gland Lesions
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ramy Refaat Ayoub Eshak, doctor, Assiut University
Other Study IDs: Major salivary gland lesions
Record Dates: First submitted 2021-11-05; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Salivary Gland Diseases
MeSH Terms: conditions — Salivary Gland Diseases | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Elastography — new dignostic tool

SUMMARY:
2.2 Aim(s) of the Research (50 words max): To investigate the diagnostic accuracy of Sonoelastography in the evaluation of major salivary gland lesions using histopathology as gold standard.

DETAILED DESCRIPTION:
Salivary gland diseases are ranging from the minor inflammatory conditions to a group of benign and malignant neoplasms. Most of the salivary gland disorders manifest themselves as the enlargement of the gland which may be associated with pain or swelling. Physical examination together with laboratory analyses may not be sufficient to discriminate these diseases . Therefore, an accurate, non invasive diagnostic method is needed to discriminate these diseases (1).

Although ultrasound-guided fine-needle aspiration cytology (FNAC) is considered the gold standard for preoperative diagnosis (2), it is an invasive method requiring significant experience to avoid complications like injury of the facial nerve as it courses within the parotid gland. This explains the continuing desire for further non-invasive diagnostic options (3).

The current imaging modalities are ultrasonography, Computed Tomography (CT) and Magnetic Resonance Imaging (MRI). Despite being highly sensitive, they lack the accuracy in differentiating benign and malignant lesions because of considerable overlap between the imaging features of benign and malignant salivary gland lesions.

Sonoelastography is a new technique that depends on the elastic properties of soft tissues, with the idea of malignant lesions being stiffer than benign or normal tissue. It may have a dependable role in diagnosing different salivary gland diseases, the same way it has been used in different parts of the body, such as the breast, lymph nodes, and thyroid (4). To the best of our knowledge, there are few studies concerning the role of elastography in the field of salivary gland disease.

ELIGIBILITY:
Inclusion Criteria

* All patients with clinically suspected lesions of parotid or submandibular glands .
* An equal number of healthy volunteers will be included during the same period as control group .

Exclusion Criteria:

• A mass with ulcerated or raw surface, involvement of the whole gland by the lesion or previous surgical treatment

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be scanned in the supine position during free-breathing, with subtle neck hyperextension and tilt to the opposite side of the evaluation. The parotid and submandibular glands will be carefully examined in the transverse and longitudinal dimensions with an 8-12 MHz linear array transducer. Doppler assessment will then be done Subsequently, sonoelastography will be performed with the same depth and focus and gained settings as for grey scale imaging. First, strain elastography will be performed. The elastogram image of the detected lesion, will be evaluated using color coding . stiffness compared to normal parenchyma using a 4-grade system like the performed. Strain ratio values of all the lesiongrading presented by Dumitriu D et al. Second, shear wave elastography will be ps ,will also be calculated individually. All will be compared with histopathology results.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
the diagnostic accuracy of Sonoelastography in the evaluation of major salivary gland lesions 2-The discrimination between different salivary gland diseases by non invasive available technique as far as possible. To investigate the dia | from october 2022 to october 2023
  Use of elastography in major salivarygland lesions benign or malignant
-The discrimination between different salivary gland diseases by non invasive available technique . -The discrimination between different salivary gland diseases by non invasive available technique as far as possible. -The discri | from october 2022 to october 2023
  Differentiation between salivary gland lesions

SECONDARY OUTCOMES:
Elastography importance in salivary gland disease | From October 2022 to October 2023
  Differentiation of Salivary gland masses

CONTACTS AND LOCATIONS:
Overall Officials: Samy abdelaziz, Principal Investigator — professor of dignostic radiology

REFERENCES:
- [Background] Dumitriu D, Dudea S, Botar-Jid C, Baciut M, Baciut G. Real-time sonoelastography of major salivary gland tumors. AJR Am J Roentgenol. 2011 Nov;197(5):W924-30. doi: 10.2214/AJR.11.6529. PMID 22021543
- [Background] Zhou H, Zhou XL, Xu HX, He YP, Bo XW, Li XL, Liu BJ, Li DD, Wang D. Initial Experience With Ultrasound Elastography for Diagnosis of Major Salivary Gland Lesions. J Ultrasound Med. 2016 Dec;35(12):2597-2606. doi: 10.7863/ultra.15.11093. Epub 2016 Oct 25. PMID 27872416
- [Background] Karaman CZ, Basak S, Polat YD, Unsal A, Taskin F, Kaya E, Gunel C. The Role of Real-Time Elastography in the Differential Diagnosis of Salivary Gland Tumors. J Ultrasound Med. 2019 Jul;38(7):1677-1683. doi: 10.1002/jum.14851. Epub 2018 Nov 13. PMID 30426518